CLINICAL TRIAL: NCT03855384
Title: Multicenter, Randomized, Double-blind, Phase Ⅲ Clinical Study to Evaluate the Efficacy and Safety of TQB2450 Plus Chemotherapy（Cisplatin or Carboplatin+ 5-Fluorouracil (5-FU) ） Versus Placebo Plus Chemotherapy as First-Line Treatment in Patients With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma（R/M SCCHN）
Brief Title: Study of TQB2450 in Patients With Recurrent or Metastatic Squamous Cell Cancer of the Head and Neck（R/M SCCHN）
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TQB2450-II-03
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-02

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450+cisplatin or carboplatin + 5-Fluorouracil (5-FU) (Experimental)
  Interventions: Drug: TQB2450+cisplatin or carboplatin + 5-Fluorouracil (5-FU)
- placebo+cisplatin or carboplatin + 5-Fluorouracil (5-FU) (Placebo Comparator)
  Interventions: Drug: placebo+cisplatin or carboplatin + 5-Fluorouracil (5-FU)

INTERVENTIONS:
Drug: TQB2450+cisplatin or carboplatin + 5-Fluorouracil (5-FU) — TQB2450 1200mg IV ，cisplatin 75 mg/m^2 IV or carboplatin AUC 5 IV on Day 1 of each week in 3-week cycles (6 cycle maximum); plus 5-FU 750 mg/m^2/day IV continuous from Day 1-5 of each 3- week cycle (6 cycle maximum).
  Arms: TQB2450+cisplatin or carboplatin + 5-Fluorouracil (5-FU)
Drug: placebo+cisplatin or carboplatin + 5-Fluorouracil (5-FU) — placebo 1200mg IV ，cisplatin 75 mg/m^2 IV or carboplatin AUC 5 IV on Day 1 of each week in 3-week cycles (6 cycle maximum); plus 5-FU 750 mg/m^2/day IV continuous from Day 1-5 of each 3- week cycle (6 cycle maximum).
  Arms: placebo+cisplatin or carboplatin + 5-Fluorouracil (5-FU)

SUMMARY:
TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed head and neck squamous cell carcinoma ，primary tumor locations of oropharynx, oral cavity, hypopharynx, or larynx.
2. No indications of local radical therapy for recurrence/metastasis head and neck squamous cell carcinoma.
3. At least one measurable lesion（ based on RECIST1.1）.
4. Can provide tissue for PD-L1 biomarker analysis: A newly obtained biopsy is preferred but an archival sample is acceptable.
5. Tumors express PD-L1,and PD-L1 expression on at least 1% of tumour cells .
6. 18 years and older.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
8. Life expectancy of at least 3 months.
9. The main organs function are normally, the following criteria are met:

   1. routine blood tests：hemoglobin（Hb）≥90g/L（no blood transfusion and blood products within 14 days）；absolute neutrophil count（ANC）≥1.5×109/L； platelets（PLT）≥100×109/L.
   2. Blood biochemical examination: alanine transaminase（ALT）and aspartate aminotransferase（AST）≤2.5×upper limit of normal (ULN)（when the liver is invaded, ALT, and AST ≤5× upper limit of normal (ULN) ）； total bilirubin (TBIL)≤1.5×upper limit of normal (ULN)（Gilbert syndrome patients，≤3×upper limit of normal (ULN)）； calculated creatinine clearance（CrCl）≥60mL/min（Creatinine clearance criteria for subjects treated with cisplatin）or CrCl≥50mL/min（Creatinine clearance criteria for subjects treated with carboplatin）(Application of Standard Cockcroft-Gault Formula).
   3. Coagulation function: activated partial thromboplastin time (aPTT) 、 international normalized ratio (INR) 、prothrombin time（PT）≤ 1.5×upper limit of normal (ULN).
   4. left ventricular ejection fraction (LVEF) measured by the Cardiac echocardiography greater than or equal to 50%.
10. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study(Such as intrauterine devices , birth control pills or condoms) ；Not Pregnant or breastfeeding women,Pregnancy before pregnancy screening（Within 7 days before the start of the study）, the women who blood / urine results were positive.
11. Understood and signed an informed consent form.

Exclusion Criteria:

1. Received systemic chemotherapy, but not chemotherapy for locally advanced disease as part of multimodality therapy (this treatment must be completed more than 6 months after informed consent).
2. Has progressive disease (PD) within six (6) months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC.
3. Prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2, anti-tumor necrosis factor CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody ,or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
4. Patients who have received cetuximab treatment within 6 moths before randomization.
5. Diagnosed and/or treated additional malignancy within 5 years prior to randomization with the exception of cured carcinoma in situ of the cervix、intramucosal carcinoma of gastrointestinal tract、breast and non-melanoma skin cancers and superficial bladder tumors.
6. Known untreated central nervous system (CNS) metastasis and/or carcinomatous meningitis. 7. Has neuropathy that is ≥ Grade 2 by Common Terminology Criteria for Adverse Events (CTCAE) version 5 criteria.

8. Previously had a severe hypersensitivity reaction to treatment with study drug or has a known sensitivity to any component of drug , including Severe hypersensitivity reaction≥3 grades (NCI CTCAEv5.0 )to monoclonal antibody 、fluorouracil、 carboplatin or cisplatin-related compounds.

9. Active autoimmune disease that may worsen with the administration of an immunostimulant. Patients with type 1 diabetes, vitiligo, psoriasis, or hypothyroidism or hyperthyroidism that do not require immunosuppression therapy are excluded.

10. Immunosuppressive drugs were used at randomization,except that:

1. Intranasal, inhaled, topical steroid or topical steroid injection (e.g. intra-articular injection)
2. Physiological doses of systemic corticosteroids (a dose of ≤ 10 mg daily prednisone (or equivalent) )
3. Preadministration of steroids for hypersensitivity reactions (e.g., preadministration of CT scans)" 11. Interstitial lung disease or non-contagious pneumonia (including past history and current illness); uncontrolled systemic diseases including diabetes, hypertension,acute lung disease, etc. except for radiotherapy-induced interstitial pneumonitis.

   12. Has any other active infection requiring systemic therapy,including patients with active tuberculosis.

   13. Unstable pleural effusion, pericardial effusion or ascites. 14. Significant cardiovascular diseases such as heart failure of New York Heart Academy(NYHA) Class 2 and above, myocardial infarction within the past 3 months, unstable arrhythmias (including QT interval ≥480 ms) or unstable Angina.

   15. Patients with immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or organ transplant history.

   16. Virological examination of hepatitis B or hepatitis C during screening meets any of the following criteria:

a. HBsAg positive and HBV DNA positive (≥1000 copies /mL); b. HCV antibody and HCV-RNA positive(The result is greater than the detection limit of the analytical method).

17. Major surgery, or unhealed wounds, ulcers or fractures within 4 weeks before randomization.

18.Has received a live-virus vaccination within 4 weeks before randomization ,allowing received seasonal flu vaccines without live viruses.

19. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of study intervention.

20. Investigator judges that the patient is not eligible to join the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
OS | up to 72 weeks
  Overall survival

SECONDARY OUTCOMES:
DOR | up to 72 weeks
  Duration of Response
PFS | up to 24 weeks
  Progression-free survival
DCR | up to 24 weeks
  Disease Control Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China